CLINICAL TRIAL: NCT04594278
Title: Remote Delivery of a Mindfulness-based Intervention to Decrease Anxiety Levels and Burnout Among Health-care Professionals During the Covid-19 Pandemic
Brief Title: COVID-19 Burnout Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-5678
Record Dates: First submitted 2020-10-18; First posted 2020-10-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Based Intervention (Experimental): A remotely delivered closed group mindfulness-based intervention using Microsoft Teams Meeting will be performed, consisting of 12-16 participants (Maximum 10 groups) and one professional with a background in mindfulness coaching . Three professionals will be coaching 2-3 groups each. The curriculum entails weekly sessions (1 hour) over a 4-week period.
  Interventions: Behavioral: Mindfulness Based Intervention

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention — A remotely delivered closed group mindfulness-based intervention using Microsoft Teams Meeting will be performed, consisting of 12-16 participants (Maximum 10 groups) and one professional with a background in mindfulness coaching . Three professionals will be coaching 2-3 groups each. The curriculum entails weekly sessions (1 hour) over a 4-week period.

SUMMARY:
The aims of this study are to assess whether the use of a MBI therapy delivered remotely is associated with a reduction of perceived stress among HCPs in the Radiation Medicine Program (RMP) and with a decrease risk of burnout during and post COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* -Employee in the radiation medicine program in UHN
* Health Care Professional (Therapist, Nurse, Physician, Resident, Physician assistant, Physician admin assistant)
* Over 18

Exclusion Criteria:

* Not working at the radiation medicine program at UHN

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | 6 months
  Perceived Stress measured by the Perceived Stress Scale/ Higher number indicates higher levels of stress. Minimum value = 10, Max Value = 40

SECONDARY OUTCOMES:
Burnout | 6 months
  Burnout assessed by the 2-item Maslach Burnout Inventory using single-item measures of emotional exhaustion and depersonalization
Coping with Stress | 6 months
  Coping measured by the BriefCOPE questionnaire. High numbers indicate that the participant is not coping well with the specific situation. Minimum value = 28, Max Value = 112

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario, Canada